CLINICAL TRIAL: NCT02768142
Title: The Impact of "Natural" Cesarean Delivery on Peripartum Maternal Blood Loss. A Randomized Controlled Trial.
Brief Title: The Impact of "Natural" Cesarean Delivery on Peripartum Maternal Blood Loss.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raed Salim (Other)
Responsible Party: Sponsor-Investigator, Raed Salim, Head of delivery unit, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00137-15-EMC
Record Dates: First submitted 2016-04-24; First posted 2016-05-11 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Natural cesarean delivery (Experimental): Placing the neonate on maternal chest immediately after the extraction from the uterus, and permitting breastfeeding during surgery.
  Interventions: Other: Natural cesarean delivery
- Standard cesarean delivery (Active Comparator): Presentation of the neonate to the mother during the operation.
  Interventions: Other: Standard cesarean delivery

INTERVENTIONS:
Other: Natural cesarean delivery — Natural cesarean delivery
  Arms: Natural cesarean delivery
Other: Standard cesarean delivery — Standard cesarean delivery
  Arms: Standard cesarean delivery

SUMMARY:
Throughout the history, the neonate was dependent on maternal touch and care for survival. In modern obstetrics, with hospital care the neonates are seldom separated from their mothers after delivery. Early skin to skin (ESTS) contact after delivery was found to increase milk production, lactation and improve maternal and neonatal outcome.

Oxytocin is the primary hormone responsible for uterine contraction and prevention of postpartum hemorrhage (PPH). ESTS contact increases oxytocin secretion.

The rate of cesarean deliveries (CDs) increased dramatically over the past decades. CD was found to decrease postpartum milk production, postpones early lactation and decreases exclusive breastfeeding.

During the typical CD, the neonate is usually presented for a short while to the mother and breastfeeding is usually delayed at least a number of hours until after the surgery and the recovery period.

Natural CD, enable ESTS contact during the surgery and give the mother the opportunity to start breastfeeding immediately after delivery of the neonate in the surgery suit. Oxytocin secretion increases with ESTS and during breastfeeding.

The aim of this study is to examine blood loss that occurs after Natural CD compared to standard CD without an ESTS contact.

ELIGIBILITY:
Inclusion Criteria:

* Estimated to be appropriate for gestational age fetus.
* Sonographic dating before 20 weeks of gestation.

Exclusion Criteria:

* Non-scheduled CD.
* Major fetal malformations.
* Multiple gestations.
* Non-controlled diabetes.
* Severe pre-eclampsia.
* General anesthesia.
* HIV carrier
* Neonatal need for early resuscitation.

Ages: 8 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Actual)
Dates: Start 2016-08; Primary Completion 2018-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level after delivery | 4 days
  Difference between pre- and post-surgical hemoglobin levels.

SECONDARY OUTCOMES:
Blood product transfusion | 4 days
  Number of Packed red blood cells and plasma products
Pain score during the operation | 1 hour
Pain score during the first day after cesarean delivery | 24 hours
  Use of analgesic drugs
Analgesia use during the operation | 1 hour
  Use of analgesic drugs
Analgesia use during the first day after cesarean delivery | 24 hours
Rate of breastfeeding at maternal hospital discharge | 4 days
Rate of breastfeeding 6 months after delivery | 6 months
Maternal satisfaction of the delivery | 4 days
  Satisfaction scale
Breast engorgement | 4 days
  Diagnosed by physical examination
Neonatal temperature after delivery | 1 hour
  Temperature

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, MD, Study Chair — Emek Medical Center, Afula, Israel
Locations (1):
- Department of Ob/Gyn, Ha'Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zafran N, Garmi G, Abdelgani S, Inbar S, Romano S, Salim R. Impact of "natural" cesarean delivery on peripartum blood loss: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jul;4(4):100642. doi: 10.1016/j.ajogmf.2022.100642. Epub 2022 Apr 8. PMID 35398585